CLINICAL TRIAL: NCT00891501
Title: The Use of Autologous Bone Marrow Mesenchymal Stem Cells in the Treatment of Articular Cartilage Defects
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Amgad Mohammed Haleem Ahmed Amin, M.B.B.S, M.Sc (Ortho), Associate Lecturer of Orthopedic Surgery, Department of Orthopedic Surgery, Cairo University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amgad
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Degenerative Arthritis; Chondral Defects; Osteochondral Defects
Keywords: autologous bone marrow mesenchymal stem cells; cartilage repair; osteoarthritis; osteochondral defects
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): Clinical case series
  Interventions: Procedure: Bone Marrow Aspiration; Procedure: Bone marrow mesenchymal stem cell implantation

INTERVENTIONS:
Procedure: Bone Marrow Aspiration — Autologous bone marrow is aspirated from the iliac crest (hip bone) of the patient using a 21-gauge bone marrow aspiration needle under complete aseptic conditions and proper anaesthesia
  Other Names: Bone marrow Biopsy
Procedure: Bone marrow mesenchymal stem cell implantation — The culture expanded mesenchymal stem cell pellet will be implanted into the osteochondral knee defect via open surgery or arthroscopically under complete sterile aseptic conditions and proper anaesthesia. The defect will be covered with an autologous periosteal flap from the proximal tibia and then sealed with human fibrin glue to seal the defect and retain the cell pellet in place
  Other Names: Autologous stem cell implantation for cartilage repair

SUMMARY:
This study is conducted to assess whether implanting autologous, culture-expanded, mesenchymal stem cells obtained from the bone marrow of patients with early osteoarthritis, cartilage defects or cartilage and underlying bone and cartilage (osteochondral) defects in joints is effective in the treatment of such conditions and alleviation of patients symptoms.

DETAILED DESCRIPTION:
All procedures are carried out after obtaining informed written consent from patients. Bone marrow is aspirated from the iliac crest (hip bone) of patients with osteochondral defects intraoperatively under complete sterile, aseptic conditions and under proper anaesthesia (general, local). The bone marrow aspirate is placed in tubes and transferred under aseptic conditions to the Tissue Culture Unit in the Biochemistry Department at the Cairo University School of Medicine where it is processed and bone marrow mesenchymal stem cells are isolated and grown in culture for 2-3 weeks. After this time interval, the cells are reprocessed and the cell pellet is obtained. Implantation of the cell pellet into the osteochondral defect of the joint after embedding it on a proper scaffold is performed followed by subsequent defect coverage with an autologous periosteal flap obtained from the proximal tibia to seal the defect and maintain the cell pellet in place. The patients will be assessed clinically with scoring systems preoperatively as well as 6 and 12 months postoperatively to assess relief of symptoms and joint function. Radiological assessment (X-rays and MRIs)of the affected joints will be performed at the same time points aforementioned to assess integrity of the formed cartilage. Second look arthroscopy and biopsy will also be performed to histologically assess the repair tissue and grade it via arthroscopic grading system according to the International Cartilage Repair Society guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Active patients (15 to 55 years).
* An isolated osteochondral defect (i.e., in a joint with an otherwise healthy articular surface - with cartilage on the opposing surface no more than grade 1 or 2 Outerbridge at the most.
* A defect that is 1 - 4 cm2 or more (up to 16 cm2).

Exclusion Criteria:

* Patients younger than 15 years and older than 55 years.
* Diffuse and advanced articular cartilage degeneration of the joint
* Axial malalignment, meniscal pathology, and ligamentous instability are RELATIVE contraindications that have to be dealt with primarily either concomitantly or before the transplantation during 1 of the 2 stages of the procedure. Refusal of the patient to address these conditions in presence of a cartilage lesion is a criterion for exclusion from the study.
* Kissing lesions (i.e., on both opposing surfaces of a joint).
* Existing infection in or around the joint & lesions of infectious or oncologic etiology.
* Debilitated patients.
* Immunocompromised patients.
* Patients with autoimmune disorders & systemic inflammatory disease.
* Preoperative poor neurological or vascular status of the affected limb.
* Specific contraindications include the use of tobacco and medications that may impair cell proliferation, such as NSAIDs and immunosuppressive drugs. Patients must be nicotine-free (stop smoking) prior to the procedure, as studies have shown that the oxidative effect of smoking impairs cell function and subsequent healing.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Clinical Scores and Radiological images | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Aziz El Singergy, M.D, Study Director — Department of Orthopedic Surgery Cairo University School of Medicine; Amgad M Haleem, M.Sc(Ortho), Principal Investigator — Department of Orthopedic Surgery Cairo University School of Medicne; Hazem M Atta, Ph.D, Study Director — Tissue Culture Unit - Department of Medical Biochemistry - Cairo University School of Medicine
Locations (1):
- Deaprtment of Orthopedic Surgery and Tissue Culture Unit of the Department of Medical Biochemistry - Cairo University School of Medicne - Kasr Al Ainy Hospitals -Al-Saray Street, El Manial, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Result] Wakitani S, Goto T, Pineda SJ, Young RG, Mansour JM, Caplan AI, Goldberg VM. Mesenchymal cell-based repair of large, full-thickness defects of articular cartilage. J Bone Joint Surg Am. 1994 Apr;76(4):579-92. doi: 10.2106/00004623-199404000-00013. PMID 8150826
- [Result] Wakitani S, Mitsuoka T, Nakamura N, Toritsuka Y, Nakamura Y, Horibe S. Autologous bone marrow stromal cell transplantation for repair of full-thickness articular cartilage defects in human patellae: two case reports. Cell Transplant. 2004;13(5):595-600. doi: 10.3727/000000004783983747. PMID 15565871
- [Result] Kuroda R, Ishida K, Matsumoto T, Akisue T, Fujioka H, Mizuno K, Ohgushi H, Wakitani S, Kurosaka M. Treatment of a full-thickness articular cartilage defect in the femoral condyle of an athlete with autologous bone-marrow stromal cells. Osteoarthritis Cartilage. 2007 Feb;15(2):226-31. doi: 10.1016/j.joca.2006.08.008. Epub 2006 Sep 26. PMID 17002893